CLINICAL TRIAL: NCT05133492
Title: A Clinical Pilot Study to Evaluate the Safety and Clinical Utility of The Nectero EAST System for Stabilization of Abdominal Aortic Aneurysms
Brief Title: First In Human Study for Small to Medium-sized Abdominal Aortic Aneurysm (AAA)
Acronym: AAA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nectero Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP001
Record Dates: First submitted 2021-11-03; First posted 2021-11-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Aortic Aneurysm; AAA; Dilation Aorta
Keywords: Abdominal Aorta; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Intervention Model Description: Population diagnosed with small to medium-sized (3.5-5.0cm) abdominal aortic aneurym.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Use of the EAST System for the stabilization treatment of AAA. The device is delivered endovascularly and placed in the AAA sac to deliver the Stabilizer Infusion Solution.
  Interventions: Device: Endovascular Aneurysm Stabilization Treatment (EAST)

INTERVENTIONS:
Device: Endovascular Aneurysm Stabilization Treatment (EAST) — Endovascular procedure: an ipsilateral ilio-femoral aortogram to confirm suitability for placement of a 14F sheath will be performed. A baseline contrast aortogram will be performed to assess vessel patency and target location of the EAST delivery catheter. Occluding and Stabilizer balloons are inflated in preparation for Stabilizer Compound delivery within the AAA sac. A post-Stabilizer angiogram will re-assess vessel patency and aorta stability. Delivery catheter is removed and discarded. The entire procedure is approximately one hour.

SUMMARY:
This is a first in human study to evaluate the safety and clinical utility of an investigational medical device called the Nectero EAST System to treat Abdominal Aortic Aneurysms or AAA.

DETAILED DESCRIPTION:
This is a Phase I multi-center, open-label study to evaluate use of the Nectero EAST system for stabilization of abdominal aortic aneurysms. Up to fifty (50) subjects will be treated at up to 10 worldwide sites with the device and followed for up to 36-months.

Primary Study Endpoints:

* Safety: absence of major events within the 1-month follow-up visit
* Success: defined as successful insertion of the delivery catheter and delivery of the Stabilizer

Secondary Study Endpoints:

* Freedom from aneurysmal sac enlargement. Enlargement is defined as diameter increase of >5mm per year, or aneurysm sac volume increase of >10% per year, as assessed by CT scans at the 1, 3, (HK only), 6, 12, 24 and 36-month follow-up visits.
* Aneurysm sac shrinkage, defined as diameter decrease of >5mm, or decrease in aneurysm sac volume of >10% as assessed by CT scans at the 1, 3 (HK only), 6, 12, 24 and 36-month follow-up visits.
* Assessment of Clinical Utility

Study duration is anticipated to be 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 years or older
* Subject can understand the purpose of the trial, voluntarily participate in the trial and sign the informed consent and is willing to complete the follow-up according to the requirements of the protocol.
* Infrarenal non-aneurysmal neck ≥15mm in length
* Aortic neck diameters ≤ 29mm
* Infrarenal neck angulation ≤ 60°
* Abdominal aneurysm from 3.5 cm to 5.0 cm.
* Overall AAA treatment length (distal renal to distal inferior margin of the aneurysm) not to exceed 10 cm
* Patient iliac or femoral arteries access vessels' size and morphology allow endovascular access of 14F introducer sheaths and catheters.
* Subject has > one-year life expectancy.
* Subject is American Society of Anesthesiology (ASA) grade 1 through 3, inclusive.
* Subject is able and willing to comply with 1, 3, 6, 12, 24 and 36-month follow-up.

Exclusion Criteria:

* Subject has an acutely ruptured or leaking or emergent aneurysm.
* Subject has a dissecting aneurysm.
* Subject has a mycotic or infected aneurysm.
* Subject has current vascular injury due to trauma.
* Subject's aneurysm is thoracic or suprarenal.
* Previous surgical or endovascular aneurysm repair for abdominal aortic aneurysm.
* Subject has thrombus, calcification, and/or plaque that may compromise delivery.
* Subject has had a myocardial infarction within six (6) months prior to enrollment.
* Subject has current angina or other active cardiac condition such as congestive heart failure, untreated or worsening atrial arrhythmia, ventricular arrhythmia, or valvular disease.
* Subject has undergone other major surgery within the 30 days prior to enrollment.
* Subjects with any transient ischemic attack (TIA) or ischemic stroke within 3 months.
* Known allergy to polyester or contrast material that cannot be pretreated.
* Subject is morbidly obese or has other clinical conditions that severely inhibit X-ray visualization of the aorta.
* Subject has connective tissue disease (e.g., Marfan syndrome, Eaton syndrome, or Bessel's disease).
* Known contraindication to undergoing angiography or anticoagulation.
* Subject has active systemic infection.
* Subject is participating in another research study.
* Subject has other medical, social, or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment and the procedures and evaluations pre- and post-treatment.
* Women of childbearing potential who are pregnant, lactating, or planning to become pregnant during the course of the trial.
* Subject has dialysis dependent renal failure or baseline serum creatinine level >2.0mg/dl.
* Subjects with liver dysfunction: alanine transaminase (ALT) or aspartate transaminase (AST) is five times higher than the normal upper limit; serum total bilirubin (STB) is two times higher than the normal upper limit.
* Subjects who are not suitable for endovascular treatment, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Procedure and Device-Related Adverse Events | Up to 30 days
  Absence of major events (procedure and device-related) within the 1-month follow-up visit
Efficacy: Successful delivery of the EAST System into the AAA sac | Up to 30 days
  Successful insertion of the delivery catheter and delivery of the Stabilizer Compound

SECONDARY OUTCOMES:
Efficacy: Evaluation of the AAA sac diameter over the 36 month follow up period. | Through study completion, an average of 3 years
  Freedom from aneurysmal sac enlargement. Enlargement is defined as diameter increase of >5mm per year, or aneurysm sac volume increase of >10% per year, as assessed by CT scans at the 1, 3, (HK only), 6, 12, 24 and 36-month follow-up visits.
Efficacy: Evaluation of the AAA sac shrinkage over the 36 month follow up period. | Through study completion, an average of 3 years
  Aneurysm sac shrinkage, defined as diameter decrease of >5mm, or decrease in aneurysm sac volume of >10% as assessed by CT scans at the 1, 3 (HK only), 6, 12, 24 and 36-month follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cheng, MD, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (5):
- Prince of Wales Private Hospital, Randwick, New South Wales, Australia
- Queen Mary Hospital, Hong Kong, Southern District, China
- Pablo Tabon Uribe Hospital, Medellín, Antioquia, Colombia
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng SWK, Eagleton M, Echeverri S, Munoz JG, Holden AH, Hill AA, Krievins D, Ramaiah V. A pilot study to evaluate a novel localized treatment to stabilize small- to medium-sized infrarenal abdominal aortic aneurysms. J Vasc Surg. 2023 Oct;78(4):929-935.e1. doi: 10.1016/j.jvs.2023.05.056. Epub 2023 Jun 15. PMID 37330148
- See also: J Vasc Surg. 2023 Jun 15:S0741-5214(23)01313-7 — https://pubmed.ncbi.nlm.nih.gov/37330148/